CLINICAL TRIAL: NCT05967377
Title: A Single Part, Open-Label, Randomised, Three-Way Crossover Study Designed to Evaluate the Pharmacokinetic Parameters and Relative Bioavailability of Sorafenib From Sorafenib (XS005) Tablets and Capsules Compared With Nexavar® (Reference Product) in Healthy Male Subjects
Brief Title: Evaluating the Pharmacokinetic Parameters and Relative Bioavailability of Sorafenib (XS005) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xspray Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: XS005-01
Record Dates: First submitted 2023-06-26; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pharmacokinetics; Bioavailability
MeSH Terms: interventions — Regimen B

STUDY DESIGN:
Intervention Model Description: Single centre, open-label, randomised, single dose, 3-way crossover comparative (PK) and bioavailability study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Sorafenib - Period 1 (Active Comparator): Subjects were admitted to the clinical unit in the morning of Day 1, and dosed with 200 mg Sorafenib (Nexavar®) in the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects remained in clinical unit until 24 h post dose (Day 2) when they were discharged from the clinical unit, and then returned to the clinical unit at 48 h and 72 h post-dose (Days 3 and 4) for a PK blood sample.The minimum washout before the next dosing period was 10 days.
  Interventions: Drug: Sorafenib - Period 1
- XS005 Sorafenib Capsule A - Period 1 (Experimental): Subjects were admitted to the clinical unit in the morning of Day 1, and dosed with 100 mg (2 x 50 mg) XS005 Sorafenib Capsule A in the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects remained in clinical unit until 24 h post dose (Day 2) when they were discharged from the clinical unit, and then returned to the clinical unit at 48 h and 72 h post-dose (Days 3 and 4) for a PK blood sample.The minimum washout before the next dosing period was 10 days.
  Interventions: Drug: XS005 Sorafenib Capsule A - Period 1
- XS005 Sorafenib Tablet A - Period 1 (Experimental): Subjects were admitted to the clinical unit in the morning of Day 1, and dosed with 100 mg XS005 Sorafenib Tablet A in the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects remained in clinical unit until 24 h post dose (Day 2) when they were discharged from the clinical unit, and then returned to the clinical unit at 48 h and 72 h post-dose (Days 3 and 4) for a PK blood sample.The minimum washout before the next dosing period was 10 days.
  Interventions: Drug: XS005 Sorafenib Tablet A - Period 1
- XS005 Sorafenib Capsule A - Period 2 (Experimental): Subjects were admitted to the clinical unit in the morning of Day 1, and dosed with 100 mg (2 x 50 mg) XS005 Sorafenib Capsule A in the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects remained in clinical unit until 24 h post dose (Day 2) when they were discharged from the clinical unit, and then returned to the clinical unit at 48 h and 72 h post-dose (Days 3 and 4) for a PK blood sample.The minimum washout before the next dosing period was 10 days.
  Interventions: Drug: XS005 Sorafenib Capsule A - Period 2
- XS005 Sorafenib Tablet A - Period 2 (Experimental): Subjects were admitted to the clinical unit in the morning of Day 1, and dosed with 100 mg XS005 Sorafenib Tablet A in the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects remained in clinical unit until 24 h post dose (Day 2) when they were discharged from the clinical unit, and then returned to the clinical unit at 48 h and 72 h post-dose (Days 3 and 4) for a PK blood sample.The minimum washout before the next dosing period was 10 days.
  Interventions: Drug: XS005 Sorafenib Tablet A - Period 2
- Sorafenib - Period 2 (Active Comparator): Subjects were admitted to the clinical unit in the morning of Day 1, and dosed with 200 mg Sorafenib (Nexavar®) in the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects remained in clinical unit until 24 h post dose (Day 2) when they were discharged from the clinical unit, and then returned to the clinical unit at 48 h and 72 h post-dose (Days 3 and 4) for a PK blood sample.The minimum washout before the next dosing period was 10 days.
  Interventions: Drug: Sorafenib - Period 2
- XS005 Sorafenib Tablet A - Period 3 (Experimental): Subjects were admitted to the clinical unit in the morning of Day 1, and dosed with 100 mg XS005 Sorafenib Tablet A in the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects remained in clinical unit until 24 h post dose (Day 2) when they were discharged from the clinical unit, and then returned to the clinical unit at 48 h and 72 h post-dose (Days 3 and 4) for a PK blood sample.The minimum washout before the next dosing period was 10 days.
  Interventions: Drug: XS005 Sorafenib Tablet A - Period 3
- Sorafenib - Period 3 (Active Comparator): Subjects were admitted to the clinical unit in the morning of Day 1, and dosed with 200 mg Sorafenib (Nexavar®) in the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects remained in clinical unit until 24 h post dose (Day 2) when they were discharged from the clinical unit, and then returned to the clinical unit at 48 h and 72 h post-dose (Days 3 and 4) for a PK blood sample.The minimum washout before the next dosing period was 10 days.
  Interventions: Drug: Sorafenib - Period 3
- XS005 Sorafenib Capsule A - Period 3 (Experimental): Subjects were admitted to the clinical unit in the morning of Day 1, and dosed with 100 mg (2 x 50 mg) XS005 Sorafenib Capsule A in the morning of Day 1 following an overnight fast of a minimum of 10 h. Subjects remained in clinical unit until 24 h post dose (Day 2) when they were discharged from the clinical unit, and then returned to the clinical unit at 48 h and 72 h post-dose (Days 3 and 4) for a PK blood sample.The minimum washout before the next dosing period was 10 days.
  Interventions: Drug: XS005 Sorafenib Capsule A - Period 3

INTERVENTIONS:
Drug: Sorafenib - Period 1 — Sorafenib (Nexavar®) Tablet, 200 mg
  Other Names: Regimen A (reference)
  Arms: Sorafenib - Period 1
Drug: XS005 Sorafenib Capsule A - Period 1 — XS005 Sorafenib Capsule A, 100 mg (2 x 50 mg)
  Other Names: Regimen B
  Arms: XS005 Sorafenib Capsule A - Period 1
Drug: XS005 Sorafenib Tablet A - Period 1 — XS005 Sorafenib Tablet A, 100 mg
  Other Names: Regimen C
  Arms: XS005 Sorafenib Tablet A - Period 1
Drug: XS005 Sorafenib Capsule A - Period 2 — XS005 Sorafenib Capsule A, 100 mg (2 x 50 mg)
  Other Names: Regimen B
  Arms: XS005 Sorafenib Capsule A - Period 2
Drug: XS005 Sorafenib Tablet A - Period 2 — XS005 Sorafenib Tablet A, 100 mg
  Other Names: Regimen C
  Arms: XS005 Sorafenib Tablet A - Period 2
Drug: Sorafenib - Period 2 — Sorafenib (Nexavar®) Tablet, 200 mg
  Other Names: Regimen A (reference)
  Arms: Sorafenib - Period 2
Drug: XS005 Sorafenib Tablet A - Period 3 — XS005 Sorafenib Tablet A, 100 mg
  Other Names: Regimen C
  Arms: XS005 Sorafenib Tablet A - Period 3
Drug: Sorafenib - Period 3 — Sorafenib (Nexavar®) Tablet, 200 mg
  Other Names: Regimen A (reference)
  Arms: Sorafenib - Period 3
Drug: XS005 Sorafenib Capsule A - Period 3 — XS005 Sorafenib Capsule A, 100 mg (2 x 50 mg)
  Other Names: Regimen B
  Arms: XS005 Sorafenib Capsule A - Period 3

SUMMARY:
This is a single centre, open-label, randomised, single dose, 3-way crossover comparative (PK) and bioavailability study in healthy male subjects comparing a 200 mg Sorafenib (Nexavar®) reference tablet (Regimen A) to XS005 Sorafenib Capsule A, 2 x 50 mg (Regimen B) and XS005 Sorafenib Tablet A,100 mg (Regimen C) formulation. It is planned to enroll 15 subjects who will receive single oral doses of investigational medicinal product (IMP) across 3 treatment periods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males.
2. Age 18 to 55 years of age.
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2.
4. Must be willing and able to communicate and participate in the whole study.
5. Must provide written informed consent.
6. Good state of health (mentally and physically) as indicated by a comprehensive clinical assessment (detailed medical history and a complete physical examination), ECG and laboratory investigations (haematology, biochemistry and urinalysis).
7. Must adhere to the contraception requirements.

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months.
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
3. Subjects who have previously been enrolled in this study.
4. History of any drug or alcohol abuse in the past 2 years.
5. Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type).
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission.
7. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
8. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening.
9. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator.
10. Subjects has amylase or lipase result exceeding >1.5 x upper limit of normal (ULN) at screening.
11. Positive drugs of abuse or alcohol breath test result.
12. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
13. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator.
14. Subject has a QT interval corrected by Fredericia (QTcF) >450 ms based on ECG at screening or at pre-dose Period 1 or a history of additional risk factors for Torsades de Pointe (eg hypokalaemia, hypomagnesia, a family history of long QT syndrome).
15. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
16. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active.
17. Donation or loss of greater than 400 mL of blood within the previous 3 months.
18. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
19. Subjects with pregnant partners.
20. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Time of Maximum Observed Plasma Concentration (Tmax) of XS005 and Nexavar® | For each study period, blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 4.
  The pharmacokinetic parameters (Tmax) were determined for the test and reference products (XS005 Sorafenib Capsule A, 2 x 50 mg and XS005 Tablet A, 100 mg and reference Sorafenib tablets (Nexavar®), respectively) for each subject using non-compartmental methods.
Maximum Observed Plasma Concentration (Cmax) of XS005 and Nexavar® | For each study period, blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 4.
  The pharmacokinetic parameters (Cmax) were determined for the test and reference products (XS005 Sorafenib Capsule A, 2 x 50 mg and XS005 Tablet A, 100 mg and reference Sorafenib tablets (Nexavar®), respectively) for each subject using non-compartmental methods.
Area Under the Plasma Concentration-Time Curve from 0 time to the last measurable of concentration AUC(0-last) of XS005 and Nexavar® | For each study period, blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 4.
  The pharmacokinetic parameters AUC(0-last) were determined for the test and reference products (XS005 Sorafenib Capsule A, 2 x 50 mg and XS005 Tablet A, 100 mg and reference Sorafenib tablets (Nexavar®), respectively) for each subject using non-compartmental methods.
Area Under the Plasma Concentration-Time Curve from 0 time Extrapolated to Infinity (AUC0-inf) of XS005 and Nexavar® | For each study period, blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 4.
  The pharmacokinetic parameters (AUC 0-inf) were determined for the test and reference products (XS005 Sorafenib Capsule A, 2 x 50 mg and XS005 Tablet A, 100 mg and reference Sorafenib tablets (Nexavar®), respectively) for each subject using non-compartmental methods.
Plasma half-life of drug (T1/2) of XS005 and Nexavar® | For each study period, blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 4.
  The pharmacokinetic parameters (T1/2) were determined for the test and reference products (XS005 Sorafenib Capsule A, 2 x 50 mg and XS005 Tablet A, 100 mg and reference Sorafenib tablets (Nexavar®), respectively) for each subject using non-compartmental methods.
Relative bioavailability (Frel) of XS005 and Nexavar® | For each study period, blood samples collected at 15 time points (including pre-dose) during the study period on Day 1 and Day 4.
  The relative bioavailability (Frel) of Sorafenib following administration of XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®).

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) (ie those beginning after dosing with study drug) | Adverse event (AE) information collected through study completion, an average of 10 weeks.
  The safety parameters TEAEs were were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
Systolic Blood Pressure (mmHg) | For each study period, Systolic Blood Pressure were collected at 4 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters Systolic Blood Pressure (mmHg) were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
Diastolic Blood Pressure (mmHg) | For each study period, Diastolic Blood Pressure were collected at 4 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters Diastolic Blood Pressure (mmHg) were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
Heart Rate (HR) (bpm) | For each study period, HR were collected at 4 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters HR summarizes were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
ECG (12-lead electrocardiogram) - Ventricular Rate (HR) (bpm) | For each study period, ECG were collected at 4 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters ECG - Ventricular Rate were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
ECG (12-lead electrocardiogram) - PR Interval (msec) | For each study period, ECG were collected at 4 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters ECG - PR Interval were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
ECG (12-lead electrocardiogram) - QRS Duration (msec) | For each study period, ECG were collected at 4 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters ECG - QRS Duration were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
ECG (12-lead electrocardiogram) - QT Interval (msec) | For each study period, ECG were collected at 4 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters ECG - QT Interval were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
ECG (12-lead electrocardiogram) - QRS Axis (°) | For each study period, ECG were collected at 4 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters ECG - QRS Axis were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
ECG (12-lead electrocardiogram) - QTcF Interval (msec) | For each study period, ECG were collected at 4 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters ECG - QTcF Interval were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics.
Number of participants with abnormal laboratory values of Clinical Chemistry | For each study period, blood samples were collected at 2 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters Clinical Chemistry were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics and presented as number of participants with abnormal laboratory values
Number of participants with abnormal hematology values | For each study period, blood samples were collected at 2 time points (including pre-dose) during the study period on Day1 and Day 2.
  The safety parameters Haematology were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics and presented as number of participants with abnormal laboratory values
Number of participants with abnormal urinalysis values | For each study period, urine samples were collected at 2 time points (including pre-dose) during the study period on Day1 and Day 2.
  The safety parameters Urinalysis were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics and presented as number of participants with abnormal laboratory values.
Number of participants with abnormal physical examination outcome | For each study period, target (symptom driven) physical examination; each subject was assessed by a physician and a physical examination was performed if the subject reported any AEs, on Day 2.
  The safety parameters physical examination outcome were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics and presented as number of subjects with abnormal physical examination outcome.
Number of participants with abnormal skin examination outcome | For each study period, skin assessments were done at 2 time points (including pre-dose) during the study period on Day 1 and Day 2.
  The safety parameters Skin assessment outcome were determined for XS005 Sorafenib Capsule A, 50 mg and Tablet A, 100 mg compared to reference Sorafenib tablets (Nexavar®) for each study subjects using descriptive statistics and presented as number of subjects with abnormal skin examination outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No